CLINICAL TRIAL: NCT02166827
Title: Effects of a NeuroAD System, for the Treatment of Alzheimer Disease: a Randomized, Double-blinded, Placebo-controlled Study
Brief Title: Effects of a NeuroAD System, for the Treatment of Alzheimer Disease
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Administrative decision
Sponsor: Neuronix Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: NRX-LT1
Record Dates: First submitted 2014-06-15; First posted 2014-06-18 (Estimated); Last update posted 2017-03-31 (Actual); Status verified 2017-03

CONDITIONS: Alzheimer's Disease
Keywords: TMS; Cognitive Stimulation; NeuroAD
MeSH Terms: conditions — Alzheimer Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- NeuroAD (Active Comparator): NeuroAd Treatment, synchronized TMS and cognitive training stimulation
  Interventions: Device: NeuroAD
- Sham TMS+Cog (Sham Comparator): Sham Device, has the same appearance and sound as the real device, combined with sham cognitive exercises. Patients come for the same number of sessions, delivers no real stimulation or cognitive training.
  Interventions: Device: Sham TMS+Cog

INTERVENTIONS:
Device: NeuroAD — Synchronized TMS and cognitive stimulation to 6 brain areas.
  Other Names: NICE
  Arms: NeuroAD
Device: Sham TMS+Cog — Sham Device, has the same appearance and sound as the real device, combined with sham cognitive exercises.
  Arms: Sham TMS+Cog

SUMMARY:
To evaluate the long-term efficacy of the NeuroAD system

DETAILED DESCRIPTION:
To evaluate the long-term efficacy of the NeuroAD system in improvement of mild- to moderate Alzheimer patients' cognitive function

ELIGIBILITY:
Main Inclusion Criteria:

1. Male or female age 60-90 years
2. Patients diagnosed with mild or moderate stage of Alzheimer's Disease, according to the DSM-IV criteria
3. MMSE score 18 to 26
4. Physical clearance for study participation as evaluated by the clinician
5. Spouse, family member or professional caregiver agree and capable of taking care for the participation of the patient in the study (answering questions regarding the patient's condition and assuming responsibility for medication)
6. Informed consent by the patient or by legally authorized person if appointed

Main Exclusion Criteria:

1. CDR 0, 0.5 or 3
2. Severe agitation
3. Mental retardation
4. History of Epileptic Seizures or Epilepsy
5. Contraindication for performing MRI scanning
6. Contraindication for receiving TMS treatment according to a TMS questionnaire
7. Patients with metal implants in the head, (i.e. cochlear implants, implanted brain stimulators and neurostimulators, aneurysm clips) with the exception of metal implants in mouth
8. Cardiac pacemakers
9. Implanted medication pumps
10. Intracardiac lines
11. Significant heart disease
12. Currently taking medication that lower the seizure threshold

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-11; Primary Completion 2015-11 (Actual); Study Completion 2015-11 (Actual)

PRIMARY OUTCOMES:
Efficacy | 3 Months
  Change from Baseline to 3 months in ADAS-Cog score and CGI-C. ADAS-Cog: Alzheimer's Disease Assessment Scale - Cognitive. CGI-C: Clinical Global Impression of Change

SECONDARY OUTCOMES:
Efficacy | 7 weeks
  Change from Baseline to week 7 in ADAS-Cog score and CGI-C. ADAS-Cog: Alzheimer's Disease Assessment Scale - Cognitive. CGI-C: Clinical Global Impression of Change
Efficacy | 6 Months
  Change from Baseline to 6 months in ADAS-Cog score and CGI-C. ADAS-Cog: Alzheimer's Disease Assessment Scale - Cognitive. CGI-C: Clinical Global Impression of Change
Efficacy | 9 Months
  Change from Baseline to 9 months in ADAS-Cog score and CGI-C. ADAS-Cog: Alzheimer's Disease Assessment Scale - Cognitive. CGI-C: Clinical Global Impression of Change

OTHER OUTCOMES:
Safety | 9 Months
  Adverse events (AE's), including serious adverse events (SAEs) occurring at any time during the trial and follow-up

CONTACTS AND LOCATIONS:
Locations (1):
- Shaare Zedek, Jerusalem, Israel

REFERENCES:
- See also: Sponsor's website — http://neuronixmedical.com/